CLINICAL TRIAL: NCT07207655
Title: The Effect of Card Game Education on the Knowledge and Health Beliefs of Hearing Impaired Individuals About Human Papillomavirus (HPV): A Randomized Controlled Trial
Brief Title: Knowledge and Beliefs of Hearing Impaired Individuals Regarding Human Papillomavirus (HPV)
Acronym: HPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sakine Yılmaz, Assistant Professor Doctor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HPV Knowledge and Beliefs
Record Dates: First submitted 2025-09-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Human Papilloma Virus (HPV); Hearing Disability
Keywords: HPV; Hearing impaired individual; health belief; health belief, information

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: control and experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Card Game Group (Experimental): HPV Card Game Group: Twenty individuals in the intervention group will receive HPV education using the card game method.
  Interventions: Other: HPV Card Game
- Control Group (No Intervention): No Intervention: Control Group Arm Description: The researcher will not apply to this group.

INTERVENTIONS:
Other: HPV Card Game — HPV Card Game Group: Twenty individuals in the intervention group will receive HPV education using the card game method.
  Arms: HPV Card Game Group

SUMMARY:
Health education is one approach to influencing individuals, groups, or communities to achieve better health. The literature indicates that increasing awareness of HPV, along with participation in early screening and vaccination programs, can positively influence attitudes and behaviors. Therefore, this research will be conducted to determine the effect of education using the card game method on the knowledge and health beliefs of hearing-impaired individuals regarding Human Papilloma Virus (HPV).

DETAILED DESCRIPTION:
Human Papillomavirus (HPV) is a highly prevalent virus worldwide, affecting both men and women. HPV is a common sexually transmitted infection that accounts for over 99% of cervical cancer cases. While HPV may not always cause cancer, screening for risky types is important. Cancer screening programs are the most important step in early cancer detection. Early diagnosis, followed by cancer screening, reduces morbidity and mortality. Access to screening services is a key factor in early cancer detection and screening. Access to information and communication with healthcare professionals are crucial for accessing cancer screening programs. Communication barriers appear to be one of the most significant barriers to early cancer diagnosis, screening, and treatment. People with hearing impairments are a unique group experiencing communication barriers. They face challenges accessing health-related information, communicating with healthcare professionals, obtaining adequate information from healthcare professionals, and understanding the information they receive. People with hearing impairments have lower literacy and health literacy rates than those without hearing impairments. Therefore, hearing-impaired individuals have less knowledge about HPV than hearing-impaired individuals, and their participation in HPV screening is more limited. It is necessary to increase the knowledge and awareness of hearing-impaired individuals about HPV screening. Health education utilizes booklets, digital instant messaging, flashcards, videos, video conferencing, and similar educational methods. One such educational method is playing with cards. Card games are fun and educational. These methods offer the advantages of being simple, playable anywhere, easy to store, suitable for children or adults in large or small groups, and actively engaging participants in the game. Studies in the literature report that providing education and information through the educational environment of the four-card game helps increase participants' knowledge and self-efficacy. Health education is one approach to influencing individuals, groups, or communities to achieve better health. The literature indicates that increasing awareness of HPV, along with participation in early screening and vaccination programs, can positively influence attitudes and behaviors. Therefore, this research will be conducted to determine the effect of education using the card game method on the knowledge and health beliefs of hearing-impaired individuals regarding Human Papilloma Virus (HPV).

ELIGIBILITY:
Inclusion Criteria:

* Participating in the study voluntarily
* Being hearing impaired
* Knowing sign language
* Being a native Turkish speaker
* Being over 18 years of age

Exclusion Criteria:

* Having a disability other than hearing loss
* Not knowing sign language
* Having a psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-28 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-test | Before the card game, individuals will be given an HPV Information Form.
  HPV Knowledge Level The HPV Information Form: The form is a short form containing 7 information statements. For each statement, 1 point is awarded for a correct answer; no points are awarded for incorrect answers or "I don't know." The total knowledge score is calculated by adding the number of correct answers. A higher score indicates a higher level of knowledge.
Pretest | Before the card game, the Health Belief Model Scale on HPV Infection and Vaccination will be administered.
  HPV Health Belief Level HPV Infection and Vaccination Health Belief Model Scale: Participant responses are scored based on item scores, and the total score for each subsection is calculated. The calculated total score is divided by the number of items in the subsection to calculate the individual's severity, barrier, susceptibility, and benefit scores. The average score for each subsection ranges from 1 to 4. A high benefit perception score indicates that a participant believes the HPV vaccine is beneficial; a high severity perception score indicates that HPV infection is a serious problem; a high barrier perception score indicates that the barriers to vaccination are numerous; and a high susceptibility perception score indicates significant sensitivity to this issue.

SECONDARY OUTCOMES:
Post-test | One month after the card game, the HPV Information Form will be applied to the individuals.
  HPV Information level The HPV Information Form: The form is a short form containing 7 information statements. For each statement, 1 point is awarded for a correct answer; no points are awarded for incorrect answers or "I don't know." The total knowledge score is calculated by adding the number of correct answers. A higher score indicates a higher level of knowledge.
Post-test | One month after the card game, the Health Belief Model Scale on HPV Infection and Vaccination will be administered.
  HPV Health Belief Model Scale HPV Infection and Vaccination Health Belief Model Scale: Participant responses are scored based on item scores, and the total score for each subsection is calculated. The calculated total score is divided by the number of items in the subsection to calculate the individual's severity, barrier, susceptibility, and benefit scores. The average score for each subsection ranges from 1 to 4. A high benefit perception score indicates that a participant believes the HPV vaccine is beneficial; a high severity perception score indicates that HPV infection is a serious problem; a high barrier perception score indicates that the barriers to vaccination are numerous; and a high susceptibility perception score indicates significant sensitivity to this issue.

CONTACTS AND LOCATIONS:
Overall Officials: Sakine Yılmaz, Assistant Professor Doctor, Principal Investigator — Çankırı Karatekin University; Bilgesu Çelik, Research assistant, Study Chair — Çankırı Karatekin University

IPD SHARING:
Plan to Share IPD: No